CLINICAL TRIAL: NCT02625389
Title: Safety and Efficacy of Lipiodol® Ultra Fluid in Association With Surgical Glues During Vascular Embolization
Brief Title: A Study to Evaluate How Safe and Effective is the Mixture of Lipiodol® Ultra Fluid and Glue When Used for Embolization Procedures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUF-44-001; CTRI/2017/05/008607 (Registry Identifier: CTRI); EUPAS15045 (Registry Identifier: EU PAS)
Record Dates: First submitted 2015-12-03; First posted 2015-12-09 (Estimated); Results first posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: Congenital Hemangioma; Hemangioendothelioma; Angiosarcoma; Arteriovenous Malformations
MeSH Terms: conditions — Hemangioendothelioma; Hemangiosarcoma; Arteriovenous Malformations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vascular embolization with Lipiodol Ultra Fluid and surgical glue (Experimental): Lipiodol Ultra Fluid (Ethyl esters of iodized fatty acids of poppy seed oil) was used in association with surgical glues.
  The glue was chosen according to the investigator and site practice and knowledge.
  The mixture ratio (Lipiodol Ultra Fluid/Glue) could vary from 20%/80% to 80%/20%.
  The volume of Lipiodol Ultra Fluid administered during the embolization procedure depended on lesion size but it should not exceed 15 mL.
  Interventions: Drug: Lipiodol Ultra Fluid with surgical glues

INTERVENTIONS:
Drug: Lipiodol Ultra Fluid with surgical glues — Lipiodol Ultra Fluid and surgical glue mixture administered via selective arterial catheterization.

SUMMARY:
This was a multicenter phase IV Post-Marketing Study. The study is designed to investigate the safety of Lipiodol® Ultra Fluid in association with surgical glues used according to each site medical practice of vascular embolization. Subjects will be enrolled with the main condition that a procedure of vascular embolization using Lipiodol® Ultra Fluid in association with surgical glues is part of their therapeutic/palliative strategy for their disease. The vascular embolization using Lipiodol® Ultra Fluid in association with surgical glue will be administered as study procedure. According to the patient need and health status a second vascular embolization using Lipiodol® Ultra Fluid in association with surgical glue may be considered by the investigator within the next 30 days after the first one. In this case, this procedure will be considered as a second study procedure. The per-procedure safety evaluation will be enabled by appropriate records of safety events during the time frame of the procedure of vascular embolization using Lipiodol® Ultra Fluid in association with surgical glues. Safety evaluation will be completed with safety records within 30 +/-3 days after the embolization procedure. Efficacy evaluation will rely on the level of lesion(s) obliteration after embolization compared to the pre-procedural target level of obliteration. Exploratory descriptive statistical methods will be used to evaluate safety and efficacy, using both the total population and subsets of subjects with similar clinical conditions.

ELIGIBILITY:
1. Female or male adult subject older than 18 years,
2. Subject presenting with vascular lesions/anomalies whether malformative (arterial, venous, arteriovenous, fistula) or tumoral (benign: hemoangioma; malignant, angiosarcoma) eligible for vascular embolization of single or multiple lesion(s), using selective transarterial catheterization and Lipiodol® Ultra Fluid in association with surgical glues as only embolization material, in the next stage of the therapeutic or palliative strategy,
3. Subject not previously treated for this/those lesion(s) by vascular embolization using Lipiodol® Ultra Fluid in association with surgical glues,
4. Subject able and willing to participate to the study,
5. Subject having read the information, having consented to audio-visual recording of informed consent process and having provided his/her consent to participate in writing by dating and signing the informed consent form or subject unable to consent in writing whose free and voluntary consent is confirmed in writing by a legal representative or impartial witness, prior to any study related procedure being conducted.

Non inclusion criteria :

1. Subject scheduled for vascular embolization using embolization materials and radiopaque material other than Lipiodol® Ultra Fluid in association with surgical glues (e.g. embolizing fluids such as alcohol or sclerosant agents; particles; implants such as coils or microcoils or balloons; powdered metals such as tantalum or tungsten), whether in combination or alone,
2. Subject with known contra-indications to vascular embolization (e.g. severe coagulation disorder, infectious syndrome),
3. Subject for whom lesion(s) to be embolized is/are acutely bleeding,
4. Subject presenting life-threatening emergency situation,
5. Subject with known contra-indication(s) to the use or with known sensitivity to Lipiodol® Ultra Fluid, to its ingredients or to drugs from a similar pharmaceutical class,
6. Subject currently treated with beta-blockers, metformin or subject who stopped beta-blockers, metformin less than 2 days prior to vascular embolization as described in Lipiodol® Ultra Fluid SmPC,
7. Subject previously treated with Interleukin II as described in Lipiodol® Ultra Fluid SmPC,
8. Subject currently treated with effective anticoagulant therapy.
9. Pregnant or breast-feeding female subject,
10. Subject having received any IMP within 7 days prior to enrolment,
11. Subject with anticipated, current or past condition (medical, psychological, social or geographical) that would compromise the subject's safety or her/his ability to participate to the study,
12. Subject unlikely to comply with the protocol, e.g. uncooperative attitude, and unlikely to complete the study,
13. Subject related to the Investigator or any other study staff or relative directly involved in the study conduct.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jing Hao, MD, Study Director — Guerbet
Locations (16):
- India (16):
  - Division of Peripheral Vascular & Endovascular sciences, Medanta-The Medicity Hospital, Gurgaon, Haryana
  - Mahatma Gandhi Missions Medical college and Hospital, Aurangabad
  - KLES Dr. Prabhakar Kore Hospital, Belagavi
  - Victoria Hospital, Bengaluru
  - Mazumdar Shaw medical Centre, Bengaluru
  - Apollo Hospital, Hyderabad
  - AIIMS, Jodhpur
  - Sanjay Gandhi Post Graduate Institute of Meducal Sciences (SGPGI), Lucknow
  - Government Medical College, Nagpur
  - BLK Super Speciality Hospital, New Delhi
  - AIIMS, New Delhi
  - B.J Govt College & Sassoon Hospitals, Pune
  - KEM Hospital, Pune
  - 7 Orange Hospitals, Pune
  - Geetanjali Medical College and Hospital, Udaipur
  - Acharya Vinobha Bhave Hospital, Wardha

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Among the 132 included subjects, 124 received the Lipiodol Ultra Fluid and surgical glue mixture and were analyzed for safety and efficacy
Groups:
- Vascular Embolization With Lipiodol Ultra Fluid and Surgical Glue: Included patients who were eligible for an embolization procedure with Lipiodol Ultra Fluid (Ethyl esters of iodized fatty acids of poppy seed oil) in association with surgical glues.
Period: Overall Study
Arm/Group | Vascular Embolization With Lipiodol Ultra Fluid and Surgical Glue
Started | 124
Completed | 124
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All patients who received the Lipiodol and surgical glue mixture
Arm/Group | Vascular Embolization With Lipiodol Ultra Fluid and Surgical Glue
Number analyzed (Participants) | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 55
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  India | 124
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 21.93 (3.49)

OUTCOME MEASURES:

1. Primary Outcome: Adverse Drug Reactions During the Embolization Procedure
Time Frame: Collected between administration of the mixture and catheterization laboratory discharge (up to 1 day)
Measure: Count of Participants; unit: Participants
Arm/Group | Vascular Embolization With Lipiodol Ultra Fluid and Surgical Glue
Number analyzed (Participants) | 124
Participants | 0

2. Secondary Outcome: Adverse Drug Reactions up to One Month After the Embolization Procedure
Time Frame: Collected between laboratory discharge and up to one month post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Vascular Embolization With Lipiodol Ultra Fluid and Surgical Glue
Number analyzed (Participants) | 124
Participants | 1

3. Secondary Outcome: Adverse Events up to One Month After the Embolization Procedure
Time Frame: Collected up to one month post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Vascular Embolization With Lipiodol Ultra Fluid and Surgical Glue
Number analyzed (Participants) | 124
Participants | 23

4. Secondary Outcome: Number of Lesions With an Actual Obliteration Score Equal to or Higher Than the Target Score
Description: Level of obliteration of the vascular bed of a lesion is evaluated in percentage (%) and distributed in a 4-level score : (1) <50%, (2) 50-75%, (3) 75-99%, and (4) 100%
Time Frame: Assessed on earliest available angiogram after the procedure (up to 30 days after the procedure)
Population: The total number of lesions treated was 138, but the actual obliteration rate was not reported for 3 lesions.
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Groups:
- First Embolization Procedure: Included patients who were eligible for an embolisation procedure with Lipiodol Ultra Fluid (Ethyl esters of iodized fatty acids of poppy seed oil) in association with surgical glues.
- Second Embolization Procedure: Included patients for whom a second embolisation procedure with Lipiodol Ultra Fluid (Ethyl esters of iodized fatty acids of poppy seed oil) in association with surgical glues was needed.
Arm/Group | First Embolization Procedure | Second Embolization Procedure
Number analyzed (Participants) | 124 | 12
Number analyzed (Lesions) | 135 | 13
Lesions | 119 | 11

ADVERSE EVENTS:
Time Frame: Adverse events were collected from informed consent signature up to one month after the last embolisation procedure (from 33 days up to 66 days after first embolisation procedure)
Arm/Group | Vascular Embolization With Lipiodol Ultra Fluid and Surgical Glue
All-Cause Mortality (participants affected / at risk) | 0/124
Serious Adverse Events (participants affected / at risk) | 2/124
Other Adverse Events (participants affected / at risk) | 23/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vascular Embolization With Lipiodol Ultra Fluid and Surgical Glue (N=124)
Hydrocephalus (Nervous system disorders) | 1 (1) — Not related to the mixture and related to the procedure
Cerebellar infarction (Nervous system disorders) | 1 (1) — Not related to the mixture and related to the procedure
Peripheral ischaemia (Vascular disorders) | 1 (1) — Not related to the mixture and related to the procedure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vascular Embolization With Lipiodol Ultra Fluid and Surgical Glue (N=124)
Injection site pain (General disorders) | 3 (3)
Pyrexia (General disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Catheter site pain (General disorders) | 1 (1)
Catheter site related reaction (General disorders) | 1 (1)
Catheter site swelling (General disorders) | 1 (1)
Injection site swelling (General disorders) | 1 (1)
Post embolisation syndrome (Injury, poisoning and procedural complications) | 6 (6)
Abdominal pain lower (Injury, poisoning and procedural complications) | 1 (1)
Constipation (Injury, poisoning and procedural complications) | 1 (1)
Dysphagia (Injury, poisoning and procedural complications) | 1 (1)
Gastritis (Injury, poisoning and procedural complications) | 1 (1)
Portal hypertensive gastropathy (Injury, poisoning and procedural complications) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1)
Dyskinesia (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 2 (2) — Related to the mixture
Blister (Skin and subcutaneous tissue disorders) | 1 (1) — Related to the mixture
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Mastication disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1)
Eye swelling (Eye disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-01-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT02625389/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT02625389/SAP_001.pdf